CLINICAL TRIAL: NCT00123786
Title: A Phase II Study of 18F-Fluorodeoxyglucose (FluGlucoScan) in Patients With Known or Suspected Soft Tissue Sarcoma
Brief Title: Study of 18F-Fluorodeoxyglucose (FluGlucoScan) in Patients With Known or Suspected Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MS-12-0009/DX-FDG-005/21933
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-03

CONDITIONS: Sarcoma
Keywords: positron emission tomography; fluorodeoxyglucose F18; tomography scanners, x-ray computed
MeSH Terms: conditions — Sarcoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Positron Emission Tomography — Positron Emission Tomography

SUMMARY:
18F-fluorodeoxyglucose (18F-FDG) has been approved by many regulatory agencies world-wide and is in widespread use in the United States, Japan and Europe. In the United States, 18F-FDG scanning in oncology is approved for federal healthcare reimbursement for non-Hodgkin's lymphoma, Hodgkin's disease, colorectal cancer, lung cancer, oesophageal cancer, melanoma, head and neck cancer and breast cancer. It has general applications in all areas where abnormal glucose metabolism may be present including in circumstances such as differentiating the tumour from scar tissue; evaluating the presence of the tumour in light of rising tumour markers and normal imaging techniques; and assessing response to therapy where other techniques are deemed to be unhelpful. Current literature suggests that functional imaging with 18F-FDG Positron Emission Tomography (PET) may play an important role in the imaging evaluation of patients with soft tissue sarcoma, including guiding biopsy; detecting local recurrence at sites of tumour resection; detecting metastatic disease; predicting and monitoring response to therapy; and assessing for prognosis. In appropriate situations, it is possibly the most effective diagnostic strategy. However, due to the low incidence of these tumours, prospective studies with large multicenter patient groups will be essential to define the exact diagnostic role of 18F-FDG PET in this clinical setting.

DETAILED DESCRIPTION:
Background: Positron Emission Tomography (PET) is a specialized nuclear medicine procedure that uses positron emitting radiolabeled tracer molecules to measure biological activity. The most common of these tracers, 18F-2-fluoro-2-deoxyglucose (FGD), an analog of glucose, is used to determine abnormal glucose metabolism in tumours and other sites. FDG has general applications where abnormal glucose metabolism may be present such as differentiating tumour from scar tissue, evaluating the presence of tumour in light of rising tumour markers and normal morphological imaging, and assessing response to therapy.

The Cross Cancer Institute has been funded to establish a PET centre and research program to prove the effectiveness of PET scanning in the Canadian health care environment and validate the data that have been developed in other jurisdictions in specific oncologic indications. A cyclotron has been installed at the Cross Cancer Institute which produces 18F-fluoride that is used in the automated synthesis of FDG. The three PET scanners in the Department of Oncologic Imaging will be used for this protocol.

Objectives:

Primary - establish the general utility and value of FDG-PET imaging in patients with known or suspected soft tissue sarcoma.

Secondary - demonstrate the safety of FDG-PET imaging by documentation of adverse events; determine whether the number of subjects available for study at the Cross Cancer Institute is sufficient to achieve statistically significant results; determine the feasibility of extending this study to a larger multicenter design.

Study Design: The proposed trial will be a Phase II, diagnostic imaging, open label, single site clinical trial. The patient population will consist of patients with known or suspected soft tissue sarcoma. This will also be a pilot study to test the feasibility of extending this trial to a larger multicenter design in view of increasing sample size and strengthening conclusions about safety and effectiveness of FDG-PET imaging in this population.

With each scan, the patient will receive a single IV injection of FDG. Initial imaging will be conducted 60 minutes after an average injection of 200-300 MBq of FDG (dose is dependent on which scanner is used and patients' weight). The images will then be examined by an experienced nuclear medicine physician and the location and intensity of abnormal FDG uptake will be reported. The referring physician will then correlate the findings with the results of clinical examinations and conventional imaging.

Statistical Analysis: The investigators will calculate the positive predictive value (PPV) of the FDG scans. They also intend to evaluate the percentage of patients in which the FDG scan outcome affected patient management.

Stopping Rules: The subject is free to withdraw at any time. The investigator also has the right to withdraw a subject from the study in the event of intercurrent illness or other reasons concerning the health or well being of the subject, or in case of lack of cooperation. Should a subject decide to withdraw or the investigator decide to withdraw the subject after administration of FDG, all efforts will be made to complete and report follow-up observations as thoroughly as possible providing consent is still valid. A complete final evaluation at the time of the subject's withdrawal is to be made with an explanation of why the subject is withdrawing or being withdrawn from the study. If the reason for withdrawing a subject from the study is a specific event or an abnormal laboratory test result, the event or test result must be recorded as an adverse event and entered into the Case Report Form.

Data Safety Monitoring Committee: Preliminary data will be analyzed for safety and effectiveness on a yearly basis until the study ends.

ELIGIBILITY:
Inclusion Criteria:

* Male or female. (If female of child bearing potential and outside of the window of 10 days since the last menstrual period, a negative serum or urine pregnancy test is required.)
* Known or suspected soft tissue sarcoma
* Age equal to or greater than 15 years
* Able and willing to follow instructions and comply with the protocol
* Provide written informed consent prior to participation in this study
* Karnofsky Performance Scale score 60-100

Exclusion Criteria:

* Nursing or pregnant females
* Age less than 15 years
* A history of malignancy other than soft-tissue sarcoma (excluding basal cell carcinoma and cervical intraepithelial neoplasia)

Recruitment: Study subjects will be referred to the Cross Cancer Oncologic Imaging Department by their physicians. The patient's study eligibility will be confirmed during the booking telephone call and eligible, interested patients will be scheduled for a PET scan.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
establish the general utility, value and clinical relevance of FDG-PET imaging in patients with known or suspected soft tissue sarcoma
demonstrate the safety of FDG-PET by documentation of adverse events

SECONDARY OUTCOMES:
determine whether the number of subjects available for study at the Cross Cancer Institute (CCI) is sufficient to achieve statistically significant results
determine the feasibility of extending this study to a larger multicenter design

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McEwan, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada